CLINICAL TRIAL: NCT00349466
Title: A Phase 2, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of Daily CF101 Administered Orally in Patients With Moderate-to-Severe Keratoconjunctivitis Sicca
Brief Title: Safety and Efficacy Study of CF101 to Treat Keratoconjunctivitis Sicca
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-201KCS
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-02

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Keratoconjunctivitis Sicca; KCS; Dry Eye
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — CF101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CF101 1mg (Experimental): CF101 1 mg given orally every 12 hours for 12 weeks
  Interventions: Drug: CF101
- Placebo (Placebo Comparator): Placebo given orally every 12 hours for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CF101 — Orally CF101 1mg
  Other Names: Piclidenoson
  Arms: CF101 1mg
Drug: Placebo — Orally matching Placebo
  Other Names: Inactive pill
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-masked, placebo-controlled, parallel-group study in adult males and females, aged 18 years and over, with a diagnosis of moderate-to-severe keratoconjunctivitis sicca (KCS). Patients will be randomized to receive either CF101 1 mg or matching placebo, given orally every 12 hours (q12h) for 12 weeks. A Screening Period of up to 4 weeks that includes a 2-week run-in period will precede a 12-week treatment period, followed by a 2-week follow-up period.

DETAILED DESCRIPTION:
At a Screening Visit, patients who provide written informed consent will have screening procedures performed, including a complete medical history, medication history, physical examination, including height, weight, sitting blood pressure, pulse rate and temperature, and clinical laboratory tests. Disease activity will be assessed using tear meniscus (TM) height, tear break-up time (BUT), fluorescein staining (FS), Schirmer test, and the Dry Eye Symptom Score (DESS). Doses of artificial tears must be stable for >2 weeks prior to the Screening Visit.

Eligible patients will begin a 2-week run-in period, during which time they will be instructed to discontinue use of all topical ophthalmic medications except for lubricant eye drops. Patients who successfully complete the 2-week run-in period will be randomized to their assigned medication (CF101 1 mg or matching placebo) to be taken orally every q12h for 12 weeks. Patients will return for assessments and a new supply of study medication at Weeks 2, 4, 8 and 12, and at Week 14 for a final follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age and over;
* Have a diagnosis of moderate-to-severe KCS as defined by: (1) Schirmer Test (ST) (without anesthesia) < 7 mm/5 min in either eye; AND (2) Positive FS, defined as a corneal punctate fluorescein staining score of ≥1 in either eye, where 0 = none and 3= severe; AND (3) At least 1 of the following ocular symptoms scored at ≥2, where 0 = none and 4 = very severe/interferes with normal activities: photophobia, blurred vision, foreign body sensation, soreness or pain, itching, burning, dryness;
* Willing to use no topical ocular treatments except for the unpreserved artificial tears;
* Doses of unpreserved artificial tears have been stable for >2 weeks prior to Screening Visit;
* Females of child-bearing potential must have a negative urine pregnancy test at screening and throughout the study, to be eligible for, and continue participation in, the study;
* Females of child-bearing potential must be willing to use 2 methods of contraception deemed adequate by the Investigator (for example oral contraceptive pills plus a barrier method) to be eligible for, and continue participation in, the study;
* Ability to complete the study in compliance with the protocol; and
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Has Sjögren's Syndrome with significant systemic non-exocrine gland involvement;
* Has Stevens-Johnson Syndrome;
* If KCS is due to rheumatoid arthritis or other autoimmune diseases, patient may not be receiving disease-modifying drugs, including methotrexate and biological agents;
* Use of systemic immunosuppressive drugs;
* Use of oral corticosteroids >10 mg prednisone, or equivalent, per day;
* Use of topical steroids within 2 weeks prior to the Screening Visit and for the duration of the study;
* Receipt of topical cyclosporine eye drops within 3 months prior to the Screening Visit and for the duration of the trial;
* Presence of chronic ocular disease other than KCS requiring topical treatment;
* Presence of post-burn ocular injury;
* Ocular herpes simplex virus infection;
* Concomitant use of contact lenses;
* Persistent intraocular inflammation or infection;
* Active blepharitis;
* Recent surgical occlusion of the lacrimal puncta;
* Subepithelial corneal scarring;
* Anesthetic or neurotrophic corneas;
* Hemoglobin level <9.0 gm/L;
* Platelet count <125,000/mm^3;
* White blood cell count <3500/mm^3;
* Serum creatinine level outside the laboratory's normal limits;
* Liver aminotransferase levels greater than 2 times the laboratory's upper limit of normal;
* Pregnancy, planned pregnancy, lactation, or inadequate contraception as judged by the Investigator;
* History of malignancy within the past 5 years (excluding basal cell carcinoma of the skin);
* Significant acute or chronic medical, ophthalmic, or psychiatric illness that, in the judgment of the Investigator, could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study;
* Participation in another investigational drug or vaccine trial concurrently or within 30 days; or
* Other conditions which would confound the study evaluations or endanger the safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irit Bareket, MD, Principal Investigator — Sheba Medical Center
Locations (3):
- Israel (3):
  - Meir Hospital, Kfar Saba
  - Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Ẕerifin

REFERENCES:
- [Result] Avni I, Garzozi HJ, Barequet IS, Segev F, Varssano D, Sartani G, Chetrit N, Bakshi E, Zadok D, Tomkins O, Litvin G, Jacobson KA, Fishman S, Harpaz Z, Farbstein M, Yehuda SB, Silverman MH, Kerns WD, Bristol DR, Cohn I, Fishman P. Treatment of dry eye syndrome with orally administered CF101: data from a phase 2 clinical trial. Ophthalmology. 2010 Jul;117(7):1287-93. doi: 10.1016/j.ophtha.2009.11.029. Epub 2010 Mar 20. PMID 20304499
- See also: Can-Fite BioPharma web site — http://www.canfite.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- CF101 1 mg: CF101 1 mg q12 hours
- Placebo: Placebo tablets q12 hours for 12 weeks
Period: Overall Study
Arm/Group | CF101 1 mg | Placebo
Started | 42 | 38
Completed | 33 | 35
Not Completed | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CF101 1 mg | Placebo | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (14.4) | 61.4 (1311.7) | 58.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 18 | 10 | 28
Region of Enrollment [Number; unit: participants]
  Israel | 42 | 38 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Schirmer Test (ST) Score in Millimeters
Description: Involved placing a standardized paper tear strip inside the lower eyelid for 5 minutes. The tear strip was then removed and the length of the strip that was wet from tears was measured in millimeters. Change from baseline is calculated. Scores range 0-35 mm, with higher scores indicating more (better) tear production.
Time Frame: 12 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Millimeters
Groups:
- CF101 1 mg; Placebo: Oral tablets given every 12 hours for 12 weeks
Arm/Group | CF101 1 mg | Placebo
Number analyzed (Participants) | 26 | 23
Millimeters | 1.25 (0.765) | 3.81 (0.814)
Statistical Analysis 1: Comparison: CF101 1 mg vs Placebo; Test type: Superiority; p = 0.027, ANCOVA

2. Primary Outcome: Change From Baseline to Week 12 in Tear Break-Up Time (BUT) in Seconds
Description: Time elapsed between a complete blink and the development of the first random dry spot on the tear film as seen under fluorescent light. Change from baseline is calculated. Scores range 0-30 seconds, with higher scores indicating better tear composition and function.
Time Frame: 12 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | CF101 1 mg | Placebo
Number analyzed (Participants) | 26 | 23
seconds | 2.83 (0.906) | 0.48 (0.083)
Statistical Analysis 1: Comparison: CF101 1 mg vs Placebo; Test type: Superiority; p = 0.083, ANCOVA

3. Primary Outcome: Number of Subjects With >25% Improvement in Fluorescein Staining of the Cornea (FS) at Week 12
Description: Severity of corneal epithelial loss as graded by Fluorescein Staining of the cornea, assessed on a 0-4+ scale with 0 = none and 4+ = severe de-epithelialization (in other words, higher scores indicate worse disease), expressed as number of participants with >25% improvement at Week 12 relative to baseline.
Time Frame: 12 weeks
Population: ITT
Measure: Number; unit: participants
Groups:
- CF101 1 mg BID; Placebo BID: Oral tablets given every 12 hours for 12 weeks
Arm/Group | CF101 1 mg BID | Placebo BID
Number analyzed (Participants) | 26 | 23
participants | 22 | 12
Statistical Analysis 1: Comparison: CF101 1 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.028, Fisher Exact

4. Secondary Outcome: Number of Subjects Experiencing Clinical Success at Week 12
Description: Proportion of subjects experiencing improvement of ≥25% over baseline at Week 12 in (a) tear breakup time (BUT), (b) superficial punctate keratitis as assessed by fluorescein staining (FS), or Schirmer Test (ST)
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | CF101 1 mg | Placebo
Number analyzed (Participants) | 26 | 23
Participants | 24 | 20
Statistical Analysis 1: Comparison: CF101 1 mg vs Placebo; Test type: Superiority; p = 0.655, Fisher Exact

5. Secondary Outcome: Change From Baseline to 12 Weeks in Dry Eye Symptom Score (DESS)
Description: DESS consists of 12 questions designed to assess the symptoms of ocular irritation, covering three areas: ocular symptoms, environmental triggers and vision-related function. Each of the 12 symptoms can be graded 0-4, with 0 indicating no symptoms over the past week, and 4 meaning constant symptoms over the past week. Scores from all answered questions are summed. The final score is multiplied by (25/number of questions answered) to give an outcome between 0 (no symptoms) to 100 (worst possible symptoms). Change from baseline is calculated.
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CF101 1 mg | Placebo
Number analyzed (Participants) | 26 | 23
score on a scale | 34.44 (25.393) | 34.53 (20.605)
Statistical Analysis 1: Comparison: CF101 1 mg vs Placebo; Test type: Superiority; p = 0.387, ANCOVA

6. Secondary Outcome: Change From Baseline to Week 12 in Tear Meniscus (TM) Height
Description: Indicator of tear volume. TM was recorded on a scale from 0-3, with 0=none, 1=trace, 2=normal, and 3=high, with higher scores meaning better tear production and integrity. Change from baseline.
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CF101 1 mg | Placebo
Number analyzed (Participants) | 26 | 23
units on a scale | 0.38 (0.637) | 0.13 (0.694)
Statistical Analysis 1: Comparison: CF101 1 mg vs Placebo; Test type: Superiority; p = 0.203, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percent Change From Baseline to Week 12 in the Use of Artificial Tears
Description: Daily use of REFRESH TEARS® Lubricant Eye Drops artificial tears supplied to each patient was recorded in diaries provided to patients. Percent change from baseline is calculated.
Time Frame: 12 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: percentage change from baseline
Arm/Group | CF101 1 mg | Placebo
Number analyzed (Participants) | 26 | 23
percentage change from baseline | 355625.0 (410162.00) | 187883.1 (477720.08)
Statistical Analysis 1: Comparison: CF101 1 mg vs Placebo; Test type: Superiority; p = .807, ANCOVA

ADVERSE EVENTS:
Time Frame: Starting on week 2 till week 12 and continue till follow up visit on week 14
Arm/Group | CF101 1 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/37
Other Adverse Events (participants affected / at risk) | 20/39 | 8/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CF101 1 mg (N=39) | Placebo (N=37)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No